CLINICAL TRIAL: NCT06160375
Title: Effect of Ultrasound-guided Erector Spine Plane Block Versus Single-injection Thoracic Paravertebral Block Via Intrathoracic Approach in Single-port Video-assisted Thoracoscopic Lung Surgeries in Postoperative Analgesia: a Randomized Controlled Trial.
Brief Title: Erector Spine Plane Block Versus Single-injection Thoracic Paravertebral Block Via Intrathoracic Approach in Single-port Video-assisted Thoracoscopic Lung Surgeries
Acronym: VAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Gaber, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pain control after VAT
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-03

CONDITIONS: Thoracoscopic Surgeries
Keywords: thoracoscopic surgery; paravertebral block; erector spine block; ultrasound guided

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (P) (Other): a scalp needle with an extended tube will be inserted into the paravertebral space at the T4 level under thoracoscopic direct vision before closing the chest. One centimeter adjacent to the vertebrae will be inserted vertically 0.5 cm under the parietal pleura with the needle, and 20 ml 0.25% bupivacaine will be injected then the field will be observed for 5 min to make sure that there is no hemorrhage or hematoma.
  Interventions: Diagnostic Test: pain assessment after video assisted thoracoscopic lung surgeries
- Group (E) (Other): the patient will be in the lateral position, by using US (Esaote MyLabSeven/ Esaote S.p.A, Genoa, Italy) a linear multifrequency 12 L probe and a 20-gauge 100 mm peripheral nerve block needle (Stimupleks Ultra 360 30°-BRA-04892510-01/B. Braun Melsungen AG, Hessen, Germany), the one-sided truncal block will be performed. The transverse process was visualized by placing the probe approximately 3 cm lateral to the spinous process of the T5 vertebrae for ESPB. When the needle advances in the craniocaudal direction with an angle of 30-40° and touched the transverse process, the presence of blood and/ or air will be checked by aspiration. Hydro-dissection was performed with 2-3 mL isotonic saline and 20 mL 0.25% bupivacaine (Marcaine 0.5%, 5 mg/mL) will be injected by observing that the erector spinae muscle (ESM) separates from the transverse process.
  Interventions: Diagnostic Test: pain assessment after video assisted thoracoscopic lung surgeries

INTERVENTIONS:
Diagnostic Test: pain assessment after video assisted thoracoscopic lung surgeries — a scalp needle with an extended tube will be inserted into the paravertebral space at the T4 level under thoracoscopic direct vision before closing the chest. One centimeter adjacent to the vertebrae will be inserted vertically 0.5 cm under the parietal pleura with the needle, and 20 ml 0.25% bupivacaine will be injected then the field will be observed for 5 min to make sure that there is no hemorrhage or hematoma.

SUMMARY:
Effect of ultrasound-guided erector spine plane block versus single-injection thoracic paravertebral block via intrathoracic approach in single-port video-assisted thoracoscopic lung surgeries in postoperative analgesia: a randomized controlled trial.

DETAILED DESCRIPTION:
Traditional thoracotomy has great trauma and severe postoperative pain. At present, thoracoscopic minimally invasive surgery is the main method of thoracic surgery. Recently, single-port video-assisted thoracoscopic (SPVAT) surgery has been widely used in thoracic surgery, especially in lung wedge resection. SPVAT lung wedge resection has the advantages of less incision, less pain, and faster recovery. It was considered to have mild postoperative pain, and ignored the need for postoperative analgesia, resulting in insufficient analgesic measures after surgery. The postoperative pain is still severe, which seriously affects the patient's postoperative recovery Pain is more than just a physical process; it is a complex, subjective phenomenon. Pain can impair the hematologic, immune, hormonal, cardiac, and respiratory systems. Pain also can limit mobility, interfere with sleep and rest, and contribute to agitation, Psychosis, aggressive behavior, and delirium. Surgical centers need to pay attention to pain management because there appears to be a direct relationship between unrelieved pain and the cost of medical care, time spent in an intensive care unit, and length of hospital stay.

Inadequate analgesia causes respiratory, hemodynamic, endocrine, and metabolic complications. The preferred drugs for postoperative pain management are opioids. Usually, morphine is used for hemodynamic stability but it has a series of side effects like nausea, vomiting, constipation, and respiratory depression. NSAIDs are also used for analgesia. It also has some side effects such as gastrointestinal disturbance, renal impairment, decreased platelet function, and impaired coagulation.

Ultrasound guidance is rapidly becoming the gold standard for regional anesthesia. There is an ever-growing weight of evidence, matched with improving technology, to show that the use of ultrasound has significant benefits. The improved safety and efficacy that ultrasound brings to regional anesthesia will help promote its use and realize the benefits that regional anesthesia has, such as decreased morbidity and mortality, superior postoperative analgesia, cost-effectiveness, decreased postoperative complications, and an improved postoperative course. Although the risk of complications is minimized with the use of ultrasound, it requires advanced experience owing to its proximity to the pleura, epidural, and subarachnoid distance.

A simpler, quicker, effective, less invasive, and less complicated analgesic method can be used for postoperative analgesia after SPVAT lung wedge resection is to inject local anesthetics (LAs) directly into the paravertebral space via the intrathoracic approach under thoracoscopic direct vision to achieve the purpose of TPB under thoracoscopic direct vision, thereby reducing postoperative pain.

The erector spine plane block (ESPB) is a new technique that is easier to visualize and perform because it is more superficial. Owing to these advantages, it has been preferred frequently for postoperative analgesia in different types of operations such as thorax, abdomen, hip, and lumbar surgeries in recent years.

.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status of I and II,
* Having body mass index (BMI) <35 kg/m2, pneumothorax, and bullae or lung nodules considered carcinoma in situ with a requirement for minimally invasive surgery and the patient will have single-port VATS.

Exclusion Criteria:

* Patient's refusal
* Age <18, pregnancy
* Spinal deformity or spinal surgical history
* Renal, hepatic patient,
* Allergies to local anesthetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative cumulative morphine consumption in the first 24 hours. | 24 hours
  postoperative cumulative morphine consumption in the first 24 hours ing

SECONDARY OUTCOMES:
1st postoperative rescue analgesic | discharge from OR to time to 1st dose of morphine
  1st dose of morphine in mg
numerical rating scale | at the PACU, 2 hours, 4 hours, 6 hours, 18 hours, and at 24 hours post operative
  pain assessment after surgery using numerical rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided